CLINICAL TRIAL: NCT05280483
Title: A Randomized, Open-label, Two-sequence, Two-cycle, Cross-over Study to Evaluate the Relative Bioavailability of ABSK021 After Single-dose Fasting and High-fat Postprandial Administration in Healthy Subjects
Brief Title: ABSK021 Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABSK021-102
Record Dates: First submitted 2022-03-07; First posted 2022-03-15 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study, a single oral dose of the tablet formulation administered under fed conditions will be compared to administration under fasted conditions to assess the effects of high-fat meal on the rate and extent of absorption and exposure.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fed states in healthy subjects (Experimental): A single 25mg dose of ABSK021 administered in a fed state.
  Interventions: Drug: ABSK021 with fed state
- Fasted states in healthy subjects (Experimental): A single 25mg dose of ABSK021 administered in a fasted state.
  Interventions: Drug: ABSK021 with fasted state

INTERVENTIONS:
Drug: ABSK021 with fed state — 25 mg ABSK021 (1x25 mg ABSK021 capsule) with food
  Arms: Fed states in healthy subjects
Drug: ABSK021 with fasted state — 25 mg ABSK021 (1x25 mg ABSK021 capsule) without food
  Arms: Fasted states in healthy subjects

SUMMARY:
This is a randomized, open-label, two-sequence, two-cycle, cross-over study to evaluate the relative bioavailability of ABSK021 after single-dose fasting and high-fat postprandial administration in healthy subjects

DETAILED DESCRIPTION:
This is a single-center, arandomized, open label, two-sequence, two-cycle, cross-over study. Up to 16 healthy subjects will be enrolled in this study. Subjects will be randomized into sequence A or sequence B (8 subjects in each study sequence), and receive single oral doses of ABSK021 on 2 occasions separated by a washout period of at least 14 days (7 half-life of ABSK021 in human). Screening will occur up to 28 days prior to the first dose. And the end of treatment visit will occur 14 days after the last dose of ABSK021.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects (male or female), age greater than or equal to 18 years and less than or equal to 45 years, single-sex subjects should no less than 4;
2. Weight ≥50 kg (≥45 kg for female), and have a body mass index (BMI) between 19 and 28 (including 19 and 28) at screening, BMI = weight (kg) / height (m) 2;
3. Physical examination, clinical laboratory examination and other related examinations are normal or acceptable deviations that are judged to be not clinically significant by the investigator;
4. Male or female subjects with child-bearing potential must agree to use effective contraception during the study and within 6 months after the administration of the last dose (see 5.4 for details), and sperm donation is not allowed for male subjects during the study; female subjects must be non-pregnant and non-lactating；pregnancy is defined as post-conception until termination of pregnancy in female， which determined by laboratory human chorionic gonadotropin (hCG) testing within 7 days prior to the first dose of this study;
5. Volunteer to participate in this study, understand the study procedures and sign the informed consent prior to any study specific procedures, good compliance and willing to follow study procedures.

Exclusion Criteria:

1. Have a history of or current cardiovascular, respiratory, hematological, hepatic, renal, gastrointestinal, endocrine, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study;
2. Have known or ongoing psychiatric disorders that would interfere with study participation as determined by the investigator;
3. Have known allergy to any drug or food;
4. Have participated in a clinical trial involving an investigational product within the last 3 months;
5. Have previously completed or withdrawn from this study or any other study investigating ABSK021, and have previously received the investigational product;
6. Have used drugs or substances that are known to be strong inhibitors or inducers of CYP3A4 within 14 days prior to the first dose (include grapefruit juice, grapefruit hybrids, pomegranates, starfruits, pomelos, Seville oranges or juice or products);
7. Have known factors that significantly affect drug absorption, distribution, metabolism, excretion, such as inability to take oral medication or significant nausea and vomiting, and malabsorption;
8. Unwilling to comply with the dietary requirements/restrictions during the study, the dietary requirements: (i) consume only the meals provided by the research center during inpatient visits, (ii) refrain from consuming strong inhibitors or inducers of CYP3A4 during the study.
9. Have an average weekly alcohol intake that exceeds 14 units within 3 months prior to screening (1 unit of alcohol is approximately 360mL of beer or 45mL of spirits with 40% alcohol content or 150mL of wine), positive for alcohol screening, or unwilling to abide by alcohol restrictions as specified in Section 5.3.3;
10. Smoking more than 5 cigarettes per day (or equivalent in tobacco or nicotine products) within 3 months prior to screening, or unwilling to abide by smoking restrictions as specified in Section 5.3.3;
11. Have a history of, in the opinion of the investigator, excessive methylxanthine/caffeine use within the previous 6 months, or unwilling to abide by restrictions as specified in Section 5.3.3. Excessive intake is defined as more than 6 units of caffeine per day; one caffeine unit is contained in 177 mL of coffee, 355 mL of tea, 355 mL of cola, or 85g of chocolate；
12. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis B e antibody (HBeAb), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody;
13. have a recent history (<45 days prior to the first dose) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection, or significantly abnormal CT examination results of chest as determined by the investigator;
14. Known history of drug abuse or have the positive results of drug abuse screening;
15. Have used or intend to use over-the-counter or prescription medication , including herbal medications, within 14 days prior to dosing and during the study;
16. Plasma donation within 30 days prior to screening or any blood donation/blood loss >500 mL during the 3 months prior to screening;
17. Have received live vaccine(s) within 2 months prior to screening, or intend to during the study;
18. The personnel involved in the planning and/or conduct of the study and their immediate family members (applies to Abbisko staff, CRO staff, and staff at the study site);
19. Abnormal vital signs, including:

    1. Ear temperature >37.5℃;
    2. Pulse>100 beats/min, or <50 beats/min;
    3. Systolic blood pressure ≥140 mmHg or <90 mmHg, diastolic blood pressure ≥90 mmHg or <50 mmHg;
20. History of gastric and intestinal surgery, or other surgical history that affects drug absorption (except appendicitis surgery);
21. Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms (female >480 ms), or family history of long QT syndrome, or have an abnormal ECG with clinical symptoms as determined by the investigator；
22. Any other clinically significant comorbidities, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-23 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Cmax | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state
AUC0-∞ | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state
AUC0-t | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state
Tmax | 4 weeks
  Pharmacokinetics parameters in fasting state and fed state

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 4 weeks
  Safety and tolerability measure by number of subjects who experience adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Shanghai, China
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China